CLINICAL TRIAL: NCT04710680
Title: Reasons for Nonattendance Inpatient Colonoscopy: a Cross-sectional Study
Brief Title: Reasons for Nonattendance Inpatient Colonoscopy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Non-IC 1.0
Record Dates: First submitted 2021-01-10; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Colonoscopy Nonattendance; Inpatient

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A
  Interventions: Other: no intervention
- group I
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The absence of colonoscopy is a clinical problem that can't be ignored. According to previous studies, the absence rate for outpatient colonoscopy is between 4% and 29%. The aim of this study is to determine the reasons for colonoscopy appointment cancellations among inpatients and to identify the factors associated with colonoscopy nonattendance.

ELIGIBILITY:
Inclusion Criteria:

* inpatients older than 18 years.
* inpatients undergoing colonoscopy

Exclusion Criteria:

* Emergency colonoscopy.
* Pregnant or breastfeeding.
* Lack of complete data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. inpatients undergoing colonoscopy.
  2. inpatients older than 18 years
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-01-30 (Estimated); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
nonattendance rate of colonoscopy appointment | 1 Day of colonoscopy
  The nonattendance rate is calculated as dividing the number of inpatients but whom colonoscopies canceled to the total number of patients multiply by 100.

SECONDARY OUTCOMES:
reason for colonoscopy cancellation | 1 Day of colonoscopy
  The root causes for colonoscopy appointment cancellation,such as patient-related reason, medical-related reason,administration-related reason,etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo First Hospital, Ningbo, Zhejiang, China